CLINICAL TRIAL: NCT06742710
Title: Liraglutide Treatment in Obese Infertile PCOS Women
Acronym: LITOP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LITOP
Record Dates: First submitted 2024-08-04; First posted 2024-12-19 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2024-12

CONDITIONS: PCOS; Obesity; Infertility
Keywords: polycystic ovary syndrome; liraglutide; infertile; obesity
MeSH Terms: conditions — Obesity; Infertility; Polycystic Ovary Syndrome | interventions — Liraglutide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Liraglutide 3.0 mg or maximum tolerable dose/day and metformin 1500 mg/day
  Interventions: Drug: Liraglutide and metformin
- Control Group (Active Comparator): Metformin 1500 mg/day
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Liraglutide and metformin — Liraglutide 3.0 mg or maximum tolerable dose/day × 12 weeks and metformin 1500 mg/day until pregnancy.
  Arms: Intervention Group
Drug: Metformin — Metformin 1500 mg/day until pregnancy
  Arms: Control Group

SUMMARY:
Liraglutide, a hypoglycemic drug, can reduce weight and improve insulin resistance while stabilizing blood glucose metabolism without increasing the risk of hypoglycemia, and has been approved by the State Food and Drug Administration of China and the US Food and Drug Administration for the treatment of obesity. Polycystic ovary syndrome (PCOS) is the main cause of female anovulatory infertility, and it is also a high-risk group of obesity. Previous studies have suggested that liraglutide improves glucose metabolism, body weight, and inflammation levels in obese women with PCOS, and improves sex hormone profiles and menstrual cycles, possibly contributing to increased fertility.

Therefore, this project intends to test the following hypothesis through a large sample randomized controlled trial in obese and infertile PCOS women who are assisted by in vitro fertilization-frozen embryo transfer (IVF-FET), using liraglutide before transplantation to reduce weight can improve the live birth rate of assisted reproduction.

ELIGIBILITY:
Inclusion Criteria:

* Women with polycystic ovary syndrome (PCOS) who meet the Rotterdam diagnostic criteria.
* Aged 20-40 years;
* 25 kg/m2 ≤ BMI ≤ 35 kg/m2;
* Have not used any anti-diabetes or weight-loss medications (metformin excluded) within the past 3 months;
* Have at least 1 transplantable frozen embryo available at the research center;
* Able to follow the study's contraceptive requirements.

Exclusion Criteria:

* Diabetic ketoacidosis or other acute complications of diabetes;
* HbA1c ≥ 9.0% before enrollment;
* Using drugs that affect appetite or nutrient absorption within the past 2 months (metformin excluded);
* Uncontrolled hyperthyroidism or hypothyroidism, hypertension, systemic autoimmune diseases, etc. that may affect pregnancy and fetal development;
* 17 hydroxyprogesterone in follicualr phase > 2.0 ng/ml;
* Serious cardiovascular, digestive, liver, or kidney diseases, HBsAg-positive chronic hepatitis B, active pulmonary tuberculosis, or AIDS, etc. that are infectious or hereditary diseases;
* Any psychiatric or psychological disorders requiring drug treatment;
* Poor pregnancy and delivery history: recurrent failed implantations ≥3 times, spontaneous abortions ≥2 times; history of stillbirth, dystocia, or birth defects; previous pregnancies with preeclampsia, eclampsia, or HELLP syndrome;
* Uncontrolled metabolic, autoimmune, or hereditary disease in the husband;
* A contraindication or relative contraindication to using GLP-1 receptor agonists (history of medullary thyroid carcinoma or family history of medullary thyroid carcinoma, acute cholecystitis or pancreatitis in the acute phase or history of previous attacks, GLP-1 receptor agonist allergy, etc.);
* Failure to comply with the contraceptive requirements of the study design;
* Failure to take medication regularly and follow up;
* Current smokers, drug addicts, alcoholics, or individuals with substance abuse;
* Participants who have participated in any clinical trial within the past 3 months prior to screening;
* Individuals with other conditions deemed unsuitable for participation in this clinical trial by the investigator;

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 890 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2029-05-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Live birth rate associated with single cycle frozen embryo transfer | At delivery
  The rate of live birth of intervention and control groups

SECONDARY OUTCOMES:
Clinical pregnancy rate of single cycle frozen embryo transfer | Thirty days after the embryo transplantation
  Viable intrauterine pregnancy confirmed by ultrasound
Incidence of newly diagnosed diabetes or gestational diabetes during pregnancy | At 28 weeks of pregnancy
  Newly diagnosed diabetes or gestational diabetes at 28 weeks of pregnancy confirmed by 75 g oral glucose tolerance test。
Pregnancy outcome and complications | From baseline to delivery
  Rate of miscarriage, multiple pregnancies, pregnancy induced hypertension, preeclampsia, HELLP syndrome, prematurity (< 37 weeks), macrosomia (birth weight > 4 kg), induction of labour, prolonged duration of labour, caesarean section, assisted delivery, peripartum increased blood loss (≥ 800 ml).
Birth weight for gestational age | At delivery
  Birth weight percentile for gestational age for neonatal sex
Apgar scores | At delivery
  Apgar scores (0~10) of the newborns at delivery
Other perinatal outcomes | At delivery
  Rate of major birth defects, stillbirth, neonatal complications, and neonatal admission to a neonatal intensive care unit.
Accumulated live birth rate | At delivery
  Accumulated liver birth rate associated with the pregnancy achieved during the first 6 months of the study
Accumulated clinical pregnancy rate | At month 6
  Accumulated clinical pregnancy rate achieved during the first 6 months of the study

OTHER OUTCOMES:
Weight | At baseline, and week 12
  Measured by the same weight scale
Oral glucose tolerance test | At baseline, week 12, 28 weeks of pregnant, six weeks after delivery
  oral glucose tolerance test was conducted to test glucose metabolism
HbA1c | At baseline and week12
  Glycosylated hemoglobin
Rate of insulin usage during pregancy | Throughout pregnancy
Number of menstrual cycles | From to 12 weeks
Free testosterone index | At baseline, week 12
  Free testosterone index
Drug-related adverse reactions | During the treatment with liraglutide or metformin
  Drug-related adverse reactions, including but not limited to, nausea, diarrhea, vomiting, decreased appetite, dyspepsia, constipation, drug allergy, hypoglycemia, acute pancreatitis, acute gallbladder disease.
Anxiety | Baseline and week 12
  Measured by Generalized Anxiety Disorder-7 scores, from 0 (no anxiety) to 21 (severe anxiety)
Depression | Baseline and week 12
  Measured by Patient Health Questionnaire-9 score from 0 (no depression) to 27 (severe depression)
Quality of life specifically for PCOS individuals | Baseline and week 12
  Measured by Modified Polycystic ovary syndrome Quality of life, with each item scores from 1 (maximum impairment) to 7 (no impairment)
Major congenital malformations | Six weeks after live birth
  Identified in the Birth Defects Prevention and Control Plan (2023-2027) issued by the National Health Commission of the People's Republic of China
Costs | At delivery
  The cost per live birth for the different intervention groups, considering both direct medical and non-medical costs, as well as indirect costs.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Obstetrics and Gynecology Hospital, Beijing
  - Haidian District Maternal and Child Health Care Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data will be available if researchers provide a methodologically sound proposal and contact to the principal investigator. Data requestors will need to sign a data access agreement.